CLINICAL TRIAL: NCT01043627
Title: Sildenafil to Tadalafil in Pulmonary Arterial Hypertension (SITAR)
Acronym: SITAR
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: United Therapeutics (Industry)
Responsible Party: Robert Frantz MD, Mayo Clinic
Other Study IDs: 09-004590
Record Dates: First submitted 2010-01-06; First posted 2010-01-07 (Estimated); Last update posted 2012-11-05 (Estimated); Status verified 2012-11

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

SUMMARY:
Assess tolerability, transition methods and clinical effects of transition from sildenafil (Revatio) to tadalafil (Adcirca) for treatment of pulmonary arterial hypertension.

DETAILED DESCRIPTION:
Sildenafil (Revatio) received approval for treatment of pulmonary arterial hypertension based upon the results of the SUPER1 study that randomized patients to sildenafil 20, 40 or 80 mg tid or matching placebo. 1 For the open label extension study, all patients received 80 mg tid. Following analysis of the data, the FDA approved 20 mg tid, indicating that "higher doses are not recommended" (Revatio PDR package insert). Although there was no significant difference between dosing groups in the overall cohort with regard to 6 minute walk, patients with idiopathic PAH did have a greater hemodynamic effect at the 80 mg tid dose, raising the possibility that the maximum approved dose was not the maximally hemodynamically effective dose for at least some patient subsets. This has resulted in a confusing situation with some clinicians treating patients with sildenafil doses substantially above the FDA recommended dose, which creates issues of cost and insurance coverage. Some patients receive up to five 20 mg Revatio (sildenafil for PH) tablets tid, increasing cost fivefold (RPFrantz, unpublished data).

Tadalafil (Adcirca) received FDA approval for treatment of PAH in May 2009, and will be available for this indication in August 2009. The pivotal Pulmonary Arterial Hypertension and Response to Tadalafil (PHIRST) study randomized 405 patients with WHO group I PAH who were either treatment naïve or on background therapy with bosentan, to receive placebo, 2.5, 10, 20 or 40 mg daily.2 A dose response was observed, with 40 mg daily meeting the primary endpoint of improvement in 6 minute walk at 16 weeks (placebo-corrected treatment effect 33 m, p < 0.01), while the composite time to clinical worsening endpoint was also met. The FDA approved dose of tadalafil for PAH is 40 mg (two 20 mg tablets) daily. 20 mg daily improved median walk distance nearly as much as the 40 mg dose, but just missed the required p value based upon the statistical plan. The PHIRST trial is the first placebo controlled trial to document an incremental benefit of phosphodiesterase-5 inhibition in patients already receiving an endothelin receptor antagonist. This has important implications for the concept of combination therapy in PAH.

Since tadalafil can be administered once daily, and the cost of the therapy is less than for sildenafil, it is anticipated that many patients will transition from sildenafil to tadalafil. The goal of this prospective and retrospective study is to gather observational data regarding how that switch is made, tolerability of the switch, and, to the extent possible with this methodology, assess clinical effects of the switch.

ELIGIBILITY:
Inclusion Criteria:

* Treatment for PAH with sildenafil at a dose of 20mg tid or greater for at least 30 days
* Clinical decision to convert from sildenafil to tadalafil therapy
* Patient consents to study participation (for patients who have already transitioned from sildenafil to tadalafil therapy prior to study initiation or identification of the patient, if the patient has provided consent for use of their medical record for research, retrospective review of the transition process will be performed. When possible, these patients will be approached about prospective data collection for the study if the transition occurred less than 3 months prior to consideration of prospective study participation)

Exclusion Criteria:

* Non-group I PAH
* Age less than 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: WHO Group I PAH patients being transitioned from sildenafil to tadalafil therapy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2009-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Describe tolerability of transition from sildenafil to tadalafil for treatment of pulmonary arterial hypertension (PAH). | 12/2011

SECONDARY OUTCOMES:
Compare Treatment Satisfaction Questionnaire for Medication (TSQM) before and 30 days (range 30-45 days) after transition and 3 months (range 12-16 weeks) after transition. | 12/2011
Compare N-terminal pro-BNP (NBNP) or brain natriuretic peptide (BNP) levels before and 3 months (range 12-16 weeks) after transition. | 12/2011
Compare 6 minute walk distance before and 3 months (range12-16 weeks) after transition. | 12/2011
Compare World Health Organization (WHO) functional class before and 3 months (range 12-16 weeks) after transition. | 12/2011
Compare echo parameters (estimated cardiac output, TAPSE, Tei index) before and 6 months (range 4-8 months) after transition. If sufficient data is available at 3 month followup, this will be compared as well. | 12/2011
Describe methods for transition from sildenafil to tadalafil for treatment of PAH. | 12/2011

CONTACTS AND LOCATIONS:
Overall Officials: Robert P Frantz, MD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Robert Bourge MD, Birmingham, Alabama
  - Ron Oudiz, Torrance, California
  - Charles Burger MD, Jacksonville, Florida

REFERENCES:
- [Derived] Frantz RP, Durst L, Burger CD, Oudiz RJ, Bourge RC, Franco V, Waxman AB, McDevitt S, Walker S. Conversion from sildenafil to tadalafil: results from the sildenafil to tadalafil in pulmonary arterial hypertension (SITAR) study. J Cardiovasc Pharmacol Ther. 2014 Nov;19(6):550-7. doi: 10.1177/1074248414528066. Epub 2014 Apr 17. PMID 24742768